CLINICAL TRIAL: NCT05714930
Title: LUPUS-BEST - Treat-to-target in Systemic Lupus Erythematosus. A Multicenter Two-armed Cluster-randomized Controlled Trial
Brief Title: LUPUS-BEST - Treat-to-target in Systemic Lupus Erythematosus
Acronym: Lupus-Best
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: University Hospital Heidelberg (Other); German Diabetes-Center, Leibniz-Institut in Düsseldorf (Other); Lupus Erythematodes-Selbsthilfegemeinschaft e.V. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUPUS-BEST
Record Dates: First submitted 2023-01-10; First posted 2023-02-06 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Treat-to-target; shared decision making
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Intervention Model Description: Multicenter, national, two-armed cluster-randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treat-to-target (Experimental): T2T will be implemented based on shared decision-making (SDM), tight control and remission as a validated treatment target (disease activity score clinical SLEDAI-2k = 0 & glucocorticoids (GC) ≤ 5 mg prednisolone equivalent & physician global assessment (PGA 0-3) < 0.5 ± immunomodulatory therapy); All intervention centers will receive T2T/SDM trainings. Patients not meeting their target criterion at study entry or at any time during the trial will be included in a tight control T2T loop of 24 weeks with assessments every 6 weeks to reach the target by adjustments of their immunomodulatory treatments. Patients in target will be assessed every 12 weeks as it is standard in clinical routine care.
  Interventions: Other: Treat-to-target as a new treatment concept
- Standard of Care (No Intervention): In the standard of care (SoC) arm, patients receive 3-to 6-monthly controls and treatment adjustments according to their physician's discretion.

INTERVENTIONS:
Other: Treat-to-target as a new treatment concept — After trial initiation, the study personnel in the intervention centers will receive a training on T2T and shared decision making (SDM). Patients in the intervention centers will receive 6-weekly visits for at least 24 weeks with therapeutic adjustments to achieve remission. In case of stable remission for 6 weeks at week 24, the patients switch to 12-weekly visits until the end of the trial at week 120. In case of flare, the patient switches to 6-weekly visits for 24 consecutive weeks. Pharmaceutical treatment decisions will be guided by current treatment standards and will be taken in accordance with SDM between patients and treating physicians.
  Arms: Treat-to-target

SUMMARY:
Multicenter, national, two-armed cluster-randomized controlled trial to evaluate the effect of a treat-to-target (T2T) strategy in in systemic lupus erythematosus (SLE). 14 centers will be randomized 1:1 to T2T or standard of care. Per arm 303 patients with SLE who are not in remission will be included and receive either tight control with 6-weekly visits with the aim to reach remission or SoC with control visits and treatment adjustment according to the physicians discretion. Study duration is 120 weeks using damage accrual and Health related Quality of Life as major outcomes.

DETAILED DESCRIPTION:
This is a multicenter, national, two-armed cluster-randomized controlled trial to evaluate the effect of a treat-to-target (T2T) strategy in in systemic lupus erythematosus (SLE) on damage progression and health related quality of life (HRQoL). The study centers will be assigned 1:1 to standard of care (SoC) or remission, defined as the absence of clinical disease activity (clinical SLEDAI =0) AND prednisolone ≤5mg/day AND physician global assessment (PGA) <0.5 on a VAS 0-3. Patient with SLE > 18 years of age who are not in remission will be eligible.

Per arm, 303 patients will be included. Intervention centers receive a standardized training on T2T and shared decision making (SDM). In the intervention centers, patients not on target enter a phase of tight control with 6-weekly visits and treatment adjustments (at least 4 visits) or until remission is reached and maintained. Patients in remission are reassessed every 12 weeks. In case of flare, they can re-enter tight control based on SDM. In the SoC arm, patients receive 3- to 6-monthly controls and treatment adjustments according to the physician's discretion. Study duration is 120 weeks using damage accrual and HRQoL as major outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with SLE according to validated classification criteria
* Age at least 18 years
* Not in a stage of remission due to

  1. Clinical SLEDAI > 0 AND/OR
  2. GC dosage above 5 mg prednisone equivalent per day AND/OR
  3. Physician global assessment ≥ 0.5 on a visual analogue scale (VAS) from 0 to 3
* Fluent German language skills
* Written informed consent

Exclusion Criteria:

* Participation in other interventional trial(s)
* Any disease or medical condition that, in the opinion of the investigator, would make the subject unsuitable for this study, would interfere with the interpretation of subject safety or study results, or is considered unsuitable by the investigator for any other reason. Examples could be:

  * Life-threatening SLE manifestations that require intensive care treatment
  * Active life-threatening diseases other than SLE
  * Active malignancies
  * Acute and chronic infections that do not allow the intensification of immunosuppressive treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Damage accrual | week 120
  Damage is defined as irreversible disease associated damage, captured by the Systemic Lupus International Collaborating Clinics/ American College of Rheumatology (SLICC/ACR-) damage index (SDI). The SDI is a validated tool to assess irreversible damage that has occurred since onset of lupus. It ranges from 0 (no damage) to 44 (highest achievable damage and worst outcome). Primary endpoint is the difference of damage accrued over 120 weeks between the two arms after 120 weeks.

SECONDARY OUTCOMES:
Health Related Quality of Life (HRQoL) | week 120
  Health related quality of life (HRGoL) is measured by the Short Form 36 questionnaire (SF-36), an established, patient-reported health survey. It contains 36 items in 8 sections. The lower the score, the higher the level of disability, "0"equalling maximum, a score of 100 no disability.
  Defined as the difference in Health Related Quality of Life between the two arms at week 120. HRQoL is measured by the disease independent Short Form 36 questionnaire (SF-36).
Disease activity reported by physicians | week 120
  Defined as the difference in Systemic Lupus Erythematodes Disease Activity Index 2000 (SLEDAI-2K) between the two arms at week 120. The SLEDAI-2K is a validated measuring tool for disease activity of SLE. Specific manifestations in 9 organ systems are evaluated. There are 24 descriptors included. 16 items are clinical, 8 are based solely on laboratory test results. They are weighted differently based on severity. The final score ranges from 0 (no disease activity) to a maximum of 105 points (highest disease activity).
Patient-reported disease activity | week 120
  Defined as the difference in Systemic Lupus Activity Questionnaire (SLAQ) between the two arms at week 120. The SLAQ asks the patient to rate disease activity on a scale of 0-10 over the past 3 months. It consists of 24 items in 9 organs/systems. Regarding disease activity, 0 is defined as no problem, 1 mild, 2 moderate and 3 severe disease activity. The respective numeric rating scale ranges from 0 = "no activity", to 10 = "most activity".
Cumulative time in remission | 120 weeks
  Remission is defined as
  * Clinical SLEDAI-2K = 0 AND
  * Physician global assessment (VAS 0-3) < 0.5 AND
  * Prednisone < 5mg/d The Systemic Lupus Erythematodes Disease Activity Index 2000 (SLEDAI-2K) is a validated measuring tool for disease activity of SLE. Specific manifestations in 9 organ systems are evaluated. There are 24 descriptors included. 16 items are clinical, 8 are based solely on laboratory test results. They are weighted differently based on severity. The final score ranges from 0 (no disease activity) to a maximum of 105 points (highest disease activity). I Physician Global Assessment is a clinical tool to assess disease activity from the clinician's perspective (rater). It is measured on a Visual Analogous Scale from 0 (no disease activity) to 3 (most severe disease activity). Assessed will be the cumulative time in remission between the two arms over 120 weeks.
Cumulative number of new organ manifestations | 120 weeks
  Defined as the difference in number of new organ manifestations according to the Systemic Lupus Erythematodes Disease Activity Index 2000 (SLEDAI-2K) between the two arms over 120 weeks. The SLEDAI-2K is a validated measuring tool for disease activity of SLE. Specific manifestations in 9 organ systems are evaluated. There are 24 descriptors included. 16 items are clinical, 8 are based solely on laboratory test results. They are weighted differently based on severity. The final score ranges from 0 (no disease activity) to a maximum of 105 points (highest disease activity).
Time to achieve remission | 120 weeks
  Defined as the mean difference in time to achieve remission defined as
  * Clinical SLEDAI-2K = 0 AND
  * Physician global assessment (VAS 0-3) < 0.5 AND
  * Prednisone < 5mg/d between the two arms over 120 weeks. The Systemic Lupus Erythematodes Disease Activity Index 2000 (SLEDAI-2K) is a validated measuring tool for disease activity of SLE. Specific manifestations in 9 organ systems are evaluated. There are 24 descriptors included. 16 items are clinical, 8 are based solely on laboratory test results. They are weighted differently based on severity. The final score ranges from 0 (no disease activity) to a maximum of 105 points (highest disease activity). Physician Global Assessment is a clinical tool to assess disease activity from the clinician's perspective (rater). It is measured on a Visual Analogous Scale from 0 (no disease activity) to 3 (most severe disease activity).
Cumulative glucocorticoid (GC) dosage at week 120 | week 120
  Difference in cumulative glucocorticoid dosage between the two arms at week 120.
Percentage of patients refusing remission as target | 120 weeks
  Defined as the difference in the percentage of patients refusing remission as target between the two arms over 120 weeks.
Percentage of physicians refusing remission as target | 120 weeks
  Defined as the difference in the percentage of physicians refusing remission as target over 120 weeks.
Drug adherence | 120 weeks
  Defined as the difference in adherence between the two arms over 120 weeks. Adherence is measured by the Medication Adherence Report Scale (MARS-5).
  MARS-5 consists of 5 items designed to reflect patient reports of nonadherence. It ranges from 5 to 25 with higher scores indicating a higher level of adherence.
Fatigue | 120 weeks
  Defined as the difference in fatigue between the two arms over 120 weeks. Fatigue is measured by the Functional Assessment of Chronic Illness Therapy (FACIT) The FACIT assesses self-reported fatigue and its impact on daily activities and function. It encompasses 13 items ranging from 0 to 52 with lower scores expressing more fatigue and lower quality of life.
Fatigue | 120 weeks
  Defined as the difference in fatigue between the two arms over 120 weeks. Fatigue is measured by the Scale and Fatigue Scale for Motor and Cognitive Functions (FSMC). The FSMC consists of 20 items on 2 subscales (cognitive and motoric fatigue) which the patient reports on a 5-point-likert scale. A maximum of 50 points can be achieved for each subscale and 100 points in total. A patient without any cognitive or motoric fatigue will achieve 20 points. ≥ points in total represent low-level of fatigue, ≥ 34 points severe fatigue.
Work productivity | 120 weeks
  Defined as the difference in work productivity between the two arms over 120 weeks. Work productivity is measured by the Work Productivity Activity Impairment Questionnaire for Lupus (WPAI:Lupus V2.0). The WPAI: Lupus V2.0 is a measurement tool for work productivity, adapted for SLE-patients. It consists of 6 items grouped in 4 domains. Outcomes for each domain are expressed as impairment percentages. Higher numbers indicate greater impairment and less productivity at work.
Evaluation of shared decision-making (SDM) by patients | 120 weeks
  Shared decision making will be assessed by the 9 item Shared Decision Making - Questionnaire (SDM-Q-9) questionnaire for patients over 120 weeks.
  The SDM-Q-9 is a patient reported questionnaire, assessing if shared decision making (SDM) occurred in the last consultation of the medical provider from the viewpoint of the patient. It consists of 2 open-ended and 9 closed questions. Each closed question is represented by a statement rated on a 6-point balanced scale ranging from 0 (= completely disagree), to 5 (= completely agree). The sum (total score) of the nine items is expressed on a scale ranging from 0 to 45. The higher the score, the greater is the level of SDM perceived.
Evaluation of shared decision-making by physicians | 120 weeks
  Shared decision making (SDM) will be assessed by the Doctor-SDM-Questionnaire (SDM-Q-Doc) for physicians over 120 weeks. The Shared decision making Q-Doc questionnaire evaluates if SDM occurred in the last consultation from the viewpoint of the physician. It is structured analogous the SDM-Q-9 and ranged from 0 to 45. The higher the score, the greater is the level of SDM perceived.
Evaluation of health utilities | 120 weeks
  The short form 6-dimensional utility index (SF-6D) is a measuring tool derived from 11 items in 6 dimensions of the Short Form -36. It ranges from = (dead) to 1 (full health).

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Schneider, MD, Principal Investigator — Heinrich-Heine University, Duesseldorf
Locations (14):
- Germany (14):
  - University Clinic Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - University Clinic Heidelberg, Heidelberg, Baden-Wurttemberg
  - University Clinic Erlangen, Erlangen, Bavaria
  - LMU Munich, Munich, Bavaria
  - University Clinic Frankfurt, Frankfurt am Main, Hesse
  - Medical University Hannover, Hanover, Lower Saxony
  - University Clinic Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Kliniken Essen Mitte, Essen, Essen, North Rhine-Westphalia
  - Rheumazentrum Ruhrgebiet Herne, Ruhr University Bochum, Herne, North Rhine-Westphalia
  - University Clinic Münster, Münster, North Rhine-Westphalia
  - University Clinic Mainz, Mainz, Rhineland-Palatinate
  - University Medical Center TU Dresden, Dresden, Saxony
  - Charité - Berlin University of Medicine, Berlin
  - UKSH Campus Kiel, Kiel